CLINICAL TRIAL: NCT05055765
Title: Comparative Evaluation Of Microneedling vs Injectable Platelet Rich Fibrin In Thin Periodontal Phenotype: A Randomised Split Mouth Clinical Trial
Brief Title: Comparative Evaluation of Microneedling and Injectable Platelet Rich Fibrin in Thin Periodontal Phenotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anjali Yadav perio
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Thin Gingiva
Keywords: periodontal phenotype
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blinding will be adopted where the investigator analysing the results will be unaware to which group the patient belongs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST GROUP I (Experimental): Thin periodontal phenotype will be treated with microneedling. A total of 4 sessions will be done with an interval of 10 days each. And all the parameters will be measured.
  Interventions: Procedure: Microneedling
- TEST GROUP II (Active Comparator): Thin periodontal phenotype will be treated with i-PRF procedure. A total of 4 sessions will be done with an interval of 10 days each. And all the parameters will be measured.
  Interventions: Procedure: injectable- platelet rich fibrin

INTERVENTIONS:
Procedure: Microneedling — MN will be carried out 1mm below of the gingival margin on the gingiva of the tooth to be treated with thirty-gauge (0.255 mm) lancet needles.
  Arms: TEST GROUP I
Procedure: injectable- platelet rich fibrin — I-PRF will be prepared according to Choukroun PRF method.
  Arms: TEST GROUP II

SUMMARY:
Evaluation of microneedling vs injectable -platelet rich fibrin on gingival phenotype in thin periodontal phenotype.

DETAILED DESCRIPTION:
INTRODUCTION The gingival phenotype and different parts of the masticatory mucosa have become the subject of considerable interest in Periodontics, especially from an aesthetic and therapeutic perspective. The periodontal phenotype has been defined as the combination of gingival phenotype and buccal bone plate thickness (bone morphotype). Gingival phenotype refers to gingival thickness (GT) and keratinized tissue width (KTW).

Gingival phenotypes can be classified as scalloped and thin or flat and thick gingiva. A gingival thickness of ≥1 mm is defined as thick phenotype and a gingival thickness of ≤1 mm as thin phenotype1. Thin gingival phenotype are very friable and might be prone to recede in response to traumatic insults, such as plaque-related inflammation and traumatic toothbrushing. Gingival recession is usually observed in the presence of trauma and inflammation in individuals with thin phenotypes, whereas pocket formation has been reported in individuals with thick phenotypes.

Soft tissue grafting in areas of thin phenotypes can enhance the quality of the gingival tissue. The best way to convert a thin soft tissue to a thick phenotype is through subepithelial connective tissue grafting Various other soft tissue augmentation procedures include: - modified roll technique and use of acellular dermal matrix. There were many drawback of these techniques such as were not cost effective, complications, second surgical site creation, healing and time consuming, etc.

Therefore marked transformation in the field of periodontics has led to the development of newer, less invasive therapeutic approaches, which allows proper management of surrounding tissues to provide best outcome of periodontal therapy. Minimally invasive treatment approaches help to achieve satisfactory therapeutic results with minimum trauma to tissues. Recent study has shown i-PRF (injectable Platelet Rich Fibrin) and Microneedling procedures to be effective in increasing gingival tissue thickness.

I-PRF prepared according to low-speed centrifugation concept can provide a significant advantage for the regeneration process, as it is rich in platelets, leucocytes and growth factors. I-PRF clots and forms a gel form after approximately 10-15 min and preserves its content in the tissue for sustained release. Recent studies have shown that in comparison to PRP and the blood clot even though there is slight or no increases in blood cell concentrations and growth factors; i- PRF was capable of inducing higher cell migration and mRNA expression of TGF- β, PDGF, osteocalcin and significant increase in type I collagen gene expression. It has been suggested that i- PRF provides a three- dimensional fibrin clot network embedding platelets, leucocytes, type I collagen, osteocalcin and growth factors acting as a dynamic gel with additional release of growth factors up to 10 days. Hence studies have documented that i-PRF results in increased gingival thickness.

Microneedling (MN) is also known as "percutaneous collagen induction therapy." Microinjuries created by MN result in minimal superficial bleedings and create a wound- healing cascade from which various growth factors, such as platelet-derived growth factors, transforming growth factors, connective tissue growth factor and fibroblast growth factors, are released. In MN, the tissue responds as if experiencing tissue trauma and the body's own collagen production is induced to preserve skin integrity. Study has shown a statistically significant increase in gingival thickness when microneedling was performed along with i- PRF in comparison to standalone i-PRF.

Only one study have evaluated effect of i-PRF alone and with microneedling on thin phenotype . To the best of our knowledge no studies have been conducted till now using microneedling alone to observe its effect on gingival thickness on thin periodontal phenotype. Considering the effects of MN and i-PRF on the biological potential, neoangiogenesis, neocollagenesis and wound, the present Randomized clinical trial is designed to compare and evaluate the effects of MN and i-PRF alone in thin periodontal phenotype. The null hypothesis is that there is no significant difference in the clinical outcome in microneedling and i-PRF on thin periodontal phenotype.

MATERIALS AND METHODOLOGY

SETTINGS: The present prospective, analytical, split mouth clinical trial will be conducted in the Department of Periodontics, Post Graduate Institute of Dental Sciences, Rohtak STUDY DESIGN: Interventional study. TIME FRAME: 12-14 months STUDY

Written and verbal consent will be taken from the willing participants. This Split mouth clinical trial will include 20 systemically healthy patients, with thin periodontal phenotype in mandibular anteriors.

Test group I : microneedling Test group II : i-PRF METHOD OF RECRUITMENT

In power analysis, it was found that a minimum of 18 cases will be required for each group at a 95% confidence level and 80% power when analysed with a mean difference of 0.5 mm and a standard deviation of 0.47 using the soft tissue thickness as a reference.

Estimating a 10% drop-out rate, the study includes 20 individuals with thin periodontal phenotypes who will consult to the Department of Periodontology, Post Graduate Institute of Dental Sciences, Rohtak .

BLINDING/MASKING Single blinding will be adopted where the investigator analysing the results will be unaware to which group the patient belongs.

PHASE I THERAPY All the participants will undergo phase-I therapy with a combination of hand scalers and curettes and ultrasonic scaler. Oral hygiene instructions will be imparted and will be reinforced at each appointment.

INTERVENTION Local anaesthesia will be administered. TEST GROUP I Thin periodontal phenotype will be treated with microneedling. A total of 4 sessions will be done with an interval of 10 days each. And all the parameters will be measured.

TEST GROUP II Thin periodontal phenotype will be treated with i-PRF procedure. A total of 4 sessions will be done with an interval of 10 days each. And all the parameters will be measured.

DATA COLLECTION METHODS To measure GT from the apical 1.5 mm of the gingival margin, a No:15 endodontic spreader with a 3-mm-diameter silicone disc will be placed in the centre and will be measured on Vernier caliper.

Keratinised tissue width will be measured with the help of UNC 15 probe with silicon disc stopper from the mucogingival junction to the free gingival margin and will be measured on Vernier caliper.

PPD will be measured using UNC 15 periodontal probe at six sites (mesiobuccal, distobuccal, mesiolingual , distolingual , and median points at buccal and lingual aspect).

GI, PI will be measured using UNC 15 periodontal probe at four sites (distofacial, mesiofacial, facial, lingual gingival margin).

All clinical parameters will be measured at baseline, 3 months and 6 months and 1 year.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution inter group comparison will be done by using Independent T test and paired t test will be use for intragroup comparison and if non-normal distributionof data, inter group comparison will be done by Mann-Whitney U test and intragroup by signed rank test. The Chi square test will be applied to analyze categoric data. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* GT of the mandibular and maxillary anterior teeth < 1 mm, gingival index (GI) of < 1
* Age 18-40 years and otherwise systemically healthy
* Patients who had completed etiological periodontal therapy with Plaque index <1, gingival index <1 and showing adequate compliance and willing to participate in the study.

Exclusion Criteria:

* Patients having systemic diseases such as hypertension, diabetes, hyperthyroidism or on medications that influence the outcome of periodontal procedure
* Pregnant and lactating women
* Smokers, tobacco users
* Previous periodontal surgery
* No haematological disorders
* Use of blood thinners
* Use of any drugs that might lead to gingival enlargement
* Stress, bruxism.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Gingival thickness (GT) | 6 months
  GT was determined at a mid-buccal location about 1mm apical to the Pocket Depth with a #15 endodontic reamer.

SECONDARY OUTCOMES:
Keratinized tissue width (KTW) | 6 months
  Keratinised tissue width will be measured with the help of UNC 15 probe with silicon disc stopper from the mucogingival junction to the free gingival margin.
Pocket Probing Depth (PD) | 6 months
  PD will be measured using UNC 15 periodontal probe at six sites (mesiobuccal, distobuccal, mesiolingual , distolingual , and median points at buccal and lingual aspect).

CONTACTS AND LOCATIONS:
Overall Officials: ANJALI YADAV, Principal Investigator — PGIDS,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India